CLINICAL TRIAL: NCT01274104
Title: A Pilot Study on the Effect of Vitamin D Treatment in Patients With Statin-Associated Myalgia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI resigned.
Sponsor: Avera McKennan Hospital & University Health Center (Other)
Responsible Party: Wael Eid, MD, Avera McKennan Hospital & University Health Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ARI-1350-Myalgia
Record Dates: First submitted 2011-01-06; First posted 2011-01-11 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Hyperlipidemia
Keywords: statin-related myalgia; high cholesterol
MeSH Terms: conditions — Hyperlipidemias; Hypercholesterolemia | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D (Active Comparator): Subjects will take 5,000 IU-capsules of vitamin D3 three times a day (for a total of 15,000 IU) for 14 days
  Interventions: Dietary Supplement: Vitamin D3
- Control (Placebo Comparator): Subjects will take 3 capsules of placebo every day for 14 days
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — 15,000 IU of Vitamin D3 every day for 14 days
  Other Names: Cholecalciferol
  Arms: Vitamin D
Other: Placebo — Placebo
  Arms: Control

SUMMARY:
The purpose of this study is to measure the effect vitamin D has in alleviating muscle pain or aches that may be caused by taking certain medications for treating high cholesterol.

DETAILED DESCRIPTION:
Participation in this study will consist of at least two study visits, expected to occur over a period of up to four weeks. Study-related medication will be provided at no cost to participants. Participants will receive either Vitamin D or placebo (sugar pill).

ELIGIBILITY:
Inclusion Criteria:

* Men and women who are between the ages of 18 and 88 years old
* A muscle symptom defined as any of the following: Myalgia (muscle aches with normal CK); Myopathy (muscle aches with increased CK up to 5 times above the upper limit of normal); or Myopathy for the purpose of further evaluation (muscle aches with increased CK up to 5 times the upper limit of normal)

Exclusion Criteria:

* Women who are pregnant, breastfeeding or planning to become pregnant
* Morbidly obese with a BMI >40 kg/m2
* Travel to southern states, areas near the Equator, etc., or use of artificial tanning beds, such that study participants have increased sunlight/UV rays exposure in the past 30 days or at any point during the trial
* Currently (within the last 2 weeks) using any of the following supplements: Vitamin D-3 (Cholecalciferol) of more than 400 IU orally daily, which would not exclude typical multi-vitamin use; Vitamin D-2 (Ergocalciferol); Calcitriol; or Coenzyme Q10
* Documented to be hyperglycemic or laboratory results show hyperglycemia prior to randomization
* Renal dysfunction defined as glomerular filtration rate less than 60 mL/min.
* Documented to have parathyroid abnormalities or parathyroid hormone laboratory results show the study participant is outside of the normal limits

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory value | 14 days
  Decrease in the level of muscle pain, based on values of Brief Pain Inventory short forms completed at the initial clinic visit and approximately four weeks later at the final clinic visit

CONTACTS AND LOCATIONS:
Overall Officials: Wael Eid, MD, Principal Investigator — Avera McKennan Hospital & University Health Center
Locations (1):
- Avera Research Institute, Sioux Falls, South Dakota, United States